CLINICAL TRIAL: NCT05033002
Title: Efficacy Testing of a Culturally Relevant Stigma Intervention With Women Living With HIV in Tanzania
Brief Title: Efficacy Testing of a Culturally Relevant Stigma Intervention With WLWH in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other); RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00109278
Record Dates: First submitted 2021-08-31; First posted 2021-09-02 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: HIV; Stigma, Social; Self Efficacy; Self Esteem; Hope; Depressive Symptoms
Keywords: HIV; women living with HIV; clinical trial; Tanzania; efficacy; feasibility
MeSH Terms: conditions — Social Stigma; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual Group (No Intervention): This group will receive treatment as usual which means that no formal stigma reduction intervention will be provided. At the end of the follow-up period, this group will be invited to view the Labda Siku Moja stigma reduction intervention without follow-up.
- Stigma Intervention Group (Experimental): This group will participate in a 5 week intervention. Each week, intervention group participants will watch one ethnodrama segment of the Labda Siku Moja stigma reduction intervention followed by a guided debrief using motivational interviewing.
  Interventions: Behavioral: Labda Siku Moja stigma reduction intervention

INTERVENTIONS:
Behavioral: Labda Siku Moja stigma reduction intervention — The Labda Siku Moja stigma reduction intervention is a tailored stigma reduction intervention for women living with HIV in Tanzania. It is comprised of five ethnodramas (video stories) culturally and linguistically relevant to the Tanzanian women living with HIV.
  Arms: Stigma Intervention Group

SUMMARY:
This study will test a stigma reduction intervention with women living with HIV in Tanzania.

DETAILED DESCRIPTION:
This study will test a culturally and linguistically relevant stigma reduction intervention, Labda Siku Moja, among women living with HIV in Tanzania.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for this study are:

* (1) women who are living with HIV;
* (2) age 18 (age of adulthood as defined by the Tanzanian government);
* (3) able and willing to voluntarily consent to participate in the study;
* (4) able to travel to a data collection in their local community (as described above);
* (5) demonstrate mental competence at time of informed consent;
* (6) verbally indicate that they plan to reside in their current community for at least 6 months after enrollment (necessary to prevent attrition);
* (7) score at the median or higher level on the Swahili Version of the Multidimensional Measure of Internalized HIV Stigma Scale.

Exclusion Criteria:

* (1) any acute psychological or physiological distress; if there is evidence of acute psychologic and/or physiologic, they will be excluded from this study and referred to an appropriate site for evaluation and treatment.
* (2) Transgender women living with HIV will not be eligible to participate in this study to reduce the potential for confounding sources of stigma recognizing that a transgender identity is highly stigmatized and culturally sensitive in Tanzania. Further, it would be exceedingly difficult to recruit a sufficient sample of transgender women living with HIV to conduct an appropriate analysis.
* (3) Participants may be enrolled in other HIV-related studies except cognitive-behavioral intervention studies addressing stigma, self-efficacy, self-esteem, and/or disclosure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael V. Relf, PhD, Principal Investigator — Duke University School of Nursing
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nyblade L, Kilonzo MN, Kisamo DH, Mtei RJ, Pan W, Relf MV. Efficacy Testing of a Culturally Relevant Stigma Reduction Intervention for Women Living With HIV in Tanzania: Protocol for a Randomized Controlled Trial. J Assoc Nurses AIDS Care. 2025 Mar 26;36(5):470-481. doi: 10.1097/JNC.0000000000000538. PMID 40138392

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment as Usual Group | Stigma Intervention Group
Started | 80 | 87
Completed | 80 | 78
Not Completed | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual Group | Stigma Intervention Group | Total
Number analyzed (Participants) | 80 | 87 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.69 (14.10) | 32.40 (12.73) | 32.54 (13.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 87 | 167
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 80 | 87 | 167
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 80 | 87 | 167
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Tanzania | 80 | 87 | 167

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Recruited as Measured by Enrollment Logs
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual Group | Stigma Intervention Group
Number analyzed (Participants) | 80 | 87
Participants | 80 | 87

2. Primary Outcome: Number of Study Participants Retained in Study as Measured by Enrollment Logs
Time Frame: 30, 90, and 180 days after intervention
Population: Analysis includes participants who completed the visit at the applicable time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual Group | Stigma Intervention Group
Number analyzed (Participants) | 80 | 87
Participants
  30 days after intervention: number analyzed (Participants) | 77 | 77
  30 days after intervention | 77 | 77
  90 days after intervention: number analyzed (Participants) | 79 | 76
  90 days after intervention | 79 | 76
  180 days after intervention: number analyzed (Participants) | 76 | 76
  180 days after intervention | 76 | 76

3. Primary Outcome: Percent of Questions Left Blank on Study Instruments
Time Frame: baseline and 30, 90, and 180 days after intervention
Population: Analysis includes participants who completed surveys at the time point indicated.
Measure: Number; unit: percent of questions left blank
Arm/Group | Treatment as Usual Group | Stigma Intervention Group
Number analyzed (Participants) | 80 | 87
percent of questions left blank
  baseline | 0 | 0
  30 days after intervention: number analyzed (Participants) | 77 | 77
  30 days after intervention | 0 | 0
  90 days after intervention: number analyzed (Participants) | 79 | 76
  90 days after intervention | 0 | 0
  180 days after intervention: number analyzed (Participants) | 76 | 76
  180 days after intervention | 0 | 0

4. Primary Outcome: Time it Takes in Minutes for Participants to Complete the Questionnaires
Time Frame: baseline and 30, 90, and 180 days after intervention
Population: Analysis includes participants who completed surveys at the time point indicated.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treatment as Usual Group | Stigma Intervention Group
Number analyzed (Participants) | 80 | 87
minutes
  Baseline | 48 (8) | 49 (8)
  30 days: number analyzed (Participants) | 77 | 77
  30 days | 42 (11) | 41 (9)
  90 days: number analyzed (Participants) | 79 | 76
  90 days | 44 (9) | 42 (8)
  180 days: number analyzed (Participants) | 76 | 76
  180 days | 43 (5) | 43 (7)

5. Primary Outcome: Number of Women Who Completed All 5 Sessions
Time Frame: up to 5 weeks
Population: This outcome measure only applies to the intervention group
Measure: Count of Participants; unit: Participants
Arm/Group | Stigma Intervention Group
Number analyzed (Participants) | 87
Participants | 76

6. Secondary Outcome: Change in Internalized Stigma, as Measured by the Swahili Version of the Multidimensional Measure of Internalized Stigma Scale
Description: Scores range from 0 to 100 with lower scores indicating less stigma and higher scores indicating more stigma
Time Frame: baseline and 30, 90, and 180 days after intervention
Population: Analysis includes participants who completed surveys at the time point indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual Group | Stigma Intervention Group
Number analyzed (Participants) | 80 | 87
score on a scale
  Baseline | 36.72 (21.59) | 40.18 (23.85)
  30 days after intervention: number analyzed (Participants) | 77 | 77
  30 days after intervention | 24.89 (19.59) | 6.01 (11.24)
  90 days after intervention: number analyzed (Participants) | 79 | 76
  90 days after intervention | 23.58 (14.92) | 5.21 (11.27)
  180 days after intervention: number analyzed (Participants) | 76 | 76
  180 days after intervention | 21.93 (13.82) | 4.61 (11.46)
Statistical Analysis 1: Comparison: Treatment as Usual Group vs Stigma Intervention Group; Test type: Superiority; p < .0001, Mixed Models Analysis — The p-value is for the t-test of the coefficient of linear (TimeXGroup) trends; Slope = -0.41 — The estimated value is for the slope of linear (TimeXGroup) trends. Controlled for significant covariates
Statistical Analysis 2: Comparison: Treatment as Usual Group vs Stigma Intervention Group; Test type: Superiority; p < .0001, Mixed Models Analysis — The p-value is for the t-test of the coefficient of quadratic (TimeXTimeXGroup) trends; Slope = 0.002 — The estimated value is for the slope of quadratic (TimeXTimeXGroup) trends. Controlled for significant covariates

7. Secondary Outcome: Change in Coping Self-efficacy, as Measured by the Swahili Version of the Coping Self-Efficacy Scale
Description: Scores range from 0 to 26, with lower scores indicating lower coping self-efficacy and higher scores indicating greater coping self-efficacy.
Time Frame: baseline and 30, 90, and 180 days after intervention
Population: Analysis includes participants who completed surveys at the time point indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual Group | Stigma Intervention Group
Number analyzed (Participants) | 80 | 87
score on a scale
  Baseline | 13.28 (4.76) | 13.17 (5.41)
  30 days after intervention: number analyzed (Participants) | 77 | 77
  30 days after intervention | 14.4 (5.63) | 17.86 (5.06)
  90 days after intervention: number analyzed (Participants) | 79 | 76
  90 days after intervention | 14.9 (5.28) | 18.00 (5.02)
  180 days after intervention: number analyzed (Participants) | 76 | 76
  180 days after intervention | 14.26 (4.49) | 17.34 (5.3)
Statistical Analysis 1: Comparison: Treatment as Usual Group vs Stigma Intervention Group; Test type: Superiority; p = .002, Mixed Models Analysis — The p-value is for the t-test of the coefficient of linear (TimeXGroup) trends; Slope = 0.06 — The estimated value is for the slope of linear (TimeXGroup) trends. Controlled for significant covariates
Statistical Analysis 2: Comparison: Treatment as Usual Group vs Stigma Intervention Group; Test type: Superiority; p = .010, Mixed Models Analysis — The p-value is for the t-test of the coefficient of quadratic (TimeXTimeXGroup) trends; Slope = -0.0003 — The estimated value is for the slope of quadratic (TimeXTimeXGroup) trends. Controlled for significant covariates

8. Secondary Outcome: Change in Self-esteem, as Measured by the Swahili Version of the Rosenberg Self-Esteem Scale
Description: Scores range from 10 to 40, with lower scores indicating lower self-esteem and higher scores indicating higher self-esteem
Time Frame: baseline and 30, 90, and 180 days after intervention
Population: Analysis includes participants who completed surveys at the time point indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual Group | Stigma Intervention Group
Number analyzed (Participants) | 80 | 87
score on a scale
  Baseline | 28.30 (4.32) | 28.17 (4.31)
  30 days after intervention: number analyzed (Participants) | 77 | 77
  30 days after intervention | 29.97 (3.69) | 32.66 (3.86)
  90 days after intervention: number analyzed (Participants) | 79 | 76
  90 days after intervention | 29.57 (4.51) | 32.26 (3.19)
  180 days after intervention: number analyzed (Participants) | 76 | 76
  180 days after intervention | 28.76 (3.31) | 32.38 (3.72)
Statistical Analysis 1: Comparison: Treatment as Usual Group vs Stigma Intervention Group; Test type: Superiority; p = .001, Mixed Models Analysis — The p-value is for the t-test of the coefficient of linear (TimeXGroup) trends; Slope = 0.05 — The estimated value is for the slope of linear (TimeXGroup) trends. Controlled for significant covariates
Statistical Analysis 2: Comparison: Treatment as Usual Group vs Stigma Intervention Group; Test type: Superiority; p = .032, Mixed Models Analysis — The p-value is for the t-test of the coefficient of quadratic (TimeXTimeXGroup) trends; Slope = -0.0002 — The estimated value is for the slope of quadratic (TimeXTimeXGroup) trends. Controlled for significant covariates

9. Secondary Outcome: Hope, as Measured by the Swahili Version of the State of Hope Scale
Description: Scores range from 6 to 24, with lower scores indicating less hope and higher scores indicating more hope
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual Group | Stigma Intervention Group
Number analyzed (Participants) | 80 | 87
score on a scale | 15.48 (3.24) | 15.82 (3.36)
Statistical Analysis 1: Comparison: Treatment as Usual Group vs Stigma Intervention Group; Test type: Superiority; p = 0.506, t-test, 2 sided; Mean Difference (Final Values) = 0.34

10. Secondary Outcome: Change in Depressive Symptoms, as Measured by the Swahili Version of the Patient Health Questionnaire 9
Description: Scores range from 0 to 27, with lower scores indicating less depressive symptoms and higher scores indicating more depressive symptoms
Time Frame: baseline and 30, 90, and 180 days after intervention
Population: Analysis includes participants who completed surveys at the time point indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual Group | Stigma Intervention Group
Number analyzed (Participants) | 80 | 87
score on a scale
  Baseline | 4.20 (3.69) | 4.63 (3.91)
  30 days after intervention: number analyzed (Participants) | 77 | 77
  30 days after intervention | 3.05 (3.69) | 2.09 (2.84)
  90 days after intervention: number analyzed (Participants) | 79 | 76
  90 days after intervention | 2.00 (2.72) | 1.77 (2.63)
  180 days after intervention: number analyzed (Participants) | 76 | 76
  180 days after intervention | 2.84 (3.51) | 1.84 (2.76)
Statistical Analysis 1: Comparison: Treatment as Usual Group vs Stigma Intervention Group; Test type: Superiority; p = .441, Mixed Models Analysis — The p-value is for the t-test of the coefficient of linear (TimeXGroup) trends; The estimated value is for the slope of linear (TimeXGroup) trends. Controlled for significant covariates
Statistical Analysis 2: Comparison: Treatment as Usual Group vs Stigma Intervention Group; Test type: Superiority; p = .734, Mixed Models Analysis — The p-value is for the t-test of the coefficient of quadratic (TimeXTimeXGroup) trends; Slope = 0.0002 — The estimated value is for the slope of quadratic (TimeXTimeXGroup) trends. Controlled for significant covariates

ADVERSE EVENTS:
Time Frame: baseline and 30, 90, and 180 days after intervention
Arm/Group | Treatment as Usual Group | Stigma Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/87
Other Adverse Events (participants affected / at risk) | 0/80 | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-23): https://cdn.clinicaltrials.gov/large-docs/02/NCT05033002/Prot_SAP_001.pdf
  • Informed Consent Form (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/02/NCT05033002/ICF_000.pdf